CLINICAL TRIAL: NCT01400555
Title: A Phase 1b Safety Study of Abiraterone Acetate (JNJ-212082) and Docetaxel in Subjects With Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Brief Title: A Safety Study of Abiraterone Acetate Administered in Combination With Docetaxel in Patients With Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Acronym: mCRPC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cougar Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR018712; COU-AA-206 (Other: Cougar Biotechnology, Inc.)
Record Dates: First submitted 2011-07-21; First posted 2011-07-22 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Prostate Neoplasms; Prostate Cancer
Keywords: Prostate Cancer; Metastatic Castration-Resistant Prostate Cancer; Abiraterone Acetate; Docetaxel; Prednisone; Dexamethasone
MeSH Terms: conditions — Prostatic Neoplasms | interventions — KPNA1 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (4):
- 001 (Experimental): Cohort 1 Docetaxel 60 mg/m2 administered once every 3 weeks + abiraterone acetate 500 mg/day + prednisone 10 mg/day
  Interventions: Drug: Cohort 1
- 002 (Experimental): Cohort 2 Docetaxel 75 mg/m2 administered once every 3 weeks + abiraterone acetate 500 mg/day + prednisone 10 mg/day
  Interventions: Drug: Cohort 2
- 003 (Experimental): Cohort 3 Docetaxel 75 mg/m2 administered once every 3 weeks + abiraterone acetate 1000 mg/day + prednisone 10 mg/day
  Interventions: Drug: Cohort 3
- 004 (Experimental): Cohort 4 Docetaxel 75 mg/m2 administered once every 3 weeks + abiraterone acetate 750 mg/day + prednisone 10 mg/day
  Interventions: Drug: Cohort 4

INTERVENTIONS:
Drug: Cohort 4 — Docetaxel 75 mg/m2 administered once every 3 weeks + abiraterone acetate 750 mg/day + prednisone 10 mg/day
  Arms: 004
Drug: Cohort 3 — Docetaxel 75 mg/m2 administered once every 3 weeks + abiraterone acetate 1000 mg/day + prednisone 10 mg/day
  Arms: 003
Drug: Cohort 2 — Docetaxel 75 mg/m2 administered once every 3 weeks + abiraterone acetate 500 mg/day + prednisone 10 mg/day
  Arms: 002
Drug: Cohort 1 — Docetaxel 60 mg/m2 administered once every 3 weeks + abiraterone acetate 500 mg/day + prednisone 10 mg/day
  Arms: 001

SUMMARY:
The purpose of this study is to evaluate the maximum safe dose of abiraterone acetate administered in combination with docetaxel plus prednisone in patients with metastatic castration-resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
This is an open-label (patients and their doctors will know the identity of study drug administered), uncontrolled (patients are not assigned to treatment by chance), multicenter safety study of escalating dose levels of abiraterone acetate administered in combination with docetaxel plus prednisone in patients with metastatic castration-resistant prostate cancer (mCRPC). This study is conducted in 2 parts. Part I consists of Screening, Treatment, assessment of dose-limiting toxicity (DLT), and determination of the maximum tolerated dose (MTD). Participants are enrolled in sequential 6-subject cohorts (groups) and administered combination therapy (abiraterone acetate and docetaxel plus prednisone) according to a dose-escalation schedule. The abiraterone acetate dose in this study will escalate from 500 mg to 1000 mg daily until the MTD is determined. The MTD is the highest combination dose among the dose combinations investigated in this study at which no more than 2 (33%) of the patients in a cohort experience a DLT. A DLT is defined by an adverse event occurring from Day 1 Week 2 (first dose of abiraterone acetate) to the day before the Day 1 Week 7 docetaxel infusion (3 weeks after the second docetaxel infusion); non-hematological toxicity >=Grade 3; Grade 4 neutropenia lasting more than 5 days, neutropenia complicated by fever, or systemic infection; thrombocytopenia <25,000/mcL, or any thrombocytopenia requiring platelet transfusion; and, any subjectively intolerable toxicity. Part II of the study consists of Continuing Treatment, when patients remain at the allocated dose level, escalate to the combination MTD, or discontinuation of docetaxel (if toxicity or intolerability develops) and continue abiraterone acetate (up to 1000 mg/day) plus prednisone, until disease progression; End of Treatment, when posttreatment efficacy and safety will be documented; and Follow-Up, when survival status and new antitumor therapy are monitored. Blood samples for pharmacokinetic and efficacy measurements will be collected at selected times during the study. Safety will be monitored. The total duration of study participation may be up to 36 months. Oral abiraterone acetate will be administered as a single daily dose (500, 750, or 1000 mg). Docetaxel will be administered once every 3 weeks as an intravenous (IV) infusion (60 or 75 mg/m2) over 1 hour. Study participants will premedicate with oral dexamethasone 8 mg 1, 3, and 12 hours before the start of each docetaxel IV infusion. Oral prednisone 5 mg will be administered twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate
* Metastatic disease documented by bone, computed tomography (CT), or magnetic resonance image (MRI) scan
* Surgical or medical castration with testosterone less than 50 ng/dL
* Prostate cancer progression documented by 1 of the following: PSA progression according to Prostate Cancer Working Group 2 (PCWG2) criteria, radiographic progression by modified Response Evaluation Criteria in Solid Tumors (RECIST) or bone scan
* Absolute neutrophil count >1,500 cells/mm3
* Platelets >100,000/µl
* Hemoglobin >=10.0 g/dL
* Eastern Cooperative Group (ECOG) status score of <=2.

Exclusion Criteria:

* Elevated liver function tests (LFTs): Serum bilirubin >upper limit of normal (ULN), alanine (ALT) or aspartate (AST) aminotransferase > 1.5 ULN concomitant with alkaline phosphatase > 2.5 ULN
* Small cell carcinoma of the prostate
* Pulmonary or brain metastasis, liver metastasis is allowed if LFTs are not elevated
* Pre-existing neuropathy or severe fluid retention
* Prior cytotoxic chemotherapy for metastatic prostate cancer
* Prior therapy with other CYP17 inhibitor(s) or investigational agent(s) targeting the androgen receptor for metastatic prostate cancer
* Treatment of primary tumor within 4 weeks of Day 1 Week 1 with surgery, radiation, chemotherapy or immunotherapy
* Use of investigational drug within 4 weeks of Day 1 Week 1 or current enrollment in an investigational drug or device study
* Prior ketoconazole for prostate cancer
* Recent history of ischemic heart disease, electrocardiogram (ECG) abnormalities, or atrial fibrillation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-09-01 (Actual); Primary Completion 2014-05-12 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a dose-limiting toxicity | Up through Week 6

SECONDARY OUTCOMES:
Proportion of patients with prostate-specific antigen (PSA) response | Up to Month 36
Time to PSA progression | Up to Month 36
Objective response rate | Up to Month 36
Radiographic progression-free survival | Up to Month 36
Survival | Up to Month 36

CONTACTS AND LOCATIONS:
Overall Officials: Cougar Biotechnology, Inc. Clinical Trial, Study Director — Cougar Biotechnology, Inc.
Locations (3):
- United States (3):
  - Los Angeles, California
  - New York, New York
  - Madison, Wisconsin

REFERENCES:
- [Derived] Huang X, Chau CH, Figg WD. Challenges to improved therapeutics for metastatic castrate resistant prostate cancer: from recent successes and failures. J Hematol Oncol. 2012 Jul 2;5:35. doi: 10.1186/1756-8722-5-35. PMID 22747660
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Phase+1b+Study+of+Abiraterone+Acetate+Plus+Prednisone+and+Docetaxel+in+Patients+with+Metastatic+Castration-resistant+Prostate+Cancer